CLINICAL TRIAL: NCT04455139
Title: A Phase II Prospective International Multicenter Clinical Trial for Eyes With Relapsed Retinoblastoma, With Randomization Depending on the Site of Relapse or on Previous Treatment
Brief Title: A Prospective International Multicenter Clinical Trial for Eyes With Relapsed Retinoblastoma
Acronym: EuRbG2018
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulties in recruiting patients due to changing in treatment standards for the target population
Sponsor: Prof. Beck Popovic Maja (Other)
Responsible Party: Sponsor-Investigator, Prof. Beck Popovic Maja, Head of pediatric hematology oncology unit, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-01967
Record Dates: First submitted 2020-04-24; First posted 2020-07-02 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Eye Cancer, Retinoblastoma
Keywords: relapsed retinoblastoma; relapse of retinoblastoma
MeSH Terms: conditions — Retinoblastoma | interventions — Topotecan; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Treatment 1a (Active Comparator): IVitC melphalan (randomized) in case of vitreous relapse only
  Interventions: Drug: Melphalan
- Treatment 1b (Experimental): IVitC topotecan (randomized) in case of vitreous relapse only
  Interventions: Drug: Topotecan
- Treatment 2a (Active Comparator): IAC melphalan (randomized) in case of retinal/diffuse subretinal relapse with no prior intra-arterial treatment
  Interventions: Drug: Melphalan
- Treatment 2b (Experimental): IAC melphalan and topotecan (randomized) in case of retinal/diffuse subretinal relapse with no prior intra-arterial treatment
  Interventions: Drug: Topotecan; Drug: Melphalan
- Treatment 2c (No Intervention): IAC melphalan and topotecan (randomized) in case of retinal/diffuse subretinal relapse with prior intra-arterial treatment
- Treatment 3a (No Intervention): sequential administration of IVitC melphalan and IAC melphalan in case of combined vitreous and retinal/diffuse subretinal relapse, if no pretreatment with intra-arterial treatment
- Treatment 3b (No Intervention): sequential administration of IVitC melphalan and IAC melphalan and topotecan, in case of combined vitreous and retinal/diffuse subretinal relapse, if prior pretreatment with intra-arterial treatment

INTERVENTIONS:
Drug: Topotecan — intravitreal or intra-arterial administration of topotecan
  Other Names: hycamtin
  Arms: Treatment 1b; Treatment 2b
Drug: Melphalan — intravitreal or intra-arterial administration of topotecan
  Other Names: alkeran
  Arms: Treatment 1a; Treatment 2a; Treatment 2b

SUMMARY:
While 95% of patients with retinoblastoma can be cured nowadays, treatment of relapse remains challenging, ending often in enucleation and/or radiotherapy. In the last 10 years, new treatment modalities have been developed to give the chance of cure also in relapse, avoiding enucleation which results in esthetic sequelae and orbital growth problems, and radiotherapy which significantly increases the risk of secondary cancers in hereditary retinoblastoma. The current protocol aims at covering all types of relapses in retinoblastoma, with treatments adapted to the site of relapse, at harmonizing the new eye- and vision-preserving treatment procedures, and evaluating their efficacy and toxicity.

DETAILED DESCRIPTION:
The study aims at improving treatment of patients with recurrent Rb through a specific approach according to the site of relapse and a uniform and well-defined treatment schedule. A precise observation of early, intermediate and long-term toxic effects with treatment recommendation will be done. For intravitreal relapse, the trial will focus on a randomization between melphalan (standard) and topotecan (investigational). For retinal / diffuse subretinal relapse in patients not having received prior IAC, it will focus on a randomization between IAC melphalan only and IAC combining melphalan+topotecan. For vitreous and retinal relapse the treatment will be a sequential administration of intravitreous and intraarterial injections (observational patients).

The duration of patient recruitment is 3 years, the duration of patient follow-up for study purposes is until at least 2 years after end of current relapse treatment. A long-term follow-up of at least 10 years on a regular basis will be proposed at the end of the study, with the aim to record the occurrence of secondary malignancies, metastases and long term sequelae.

The overall objective is to provide a conservative eye-preserving treatment for pediatric patients with Rb who have failed prior standard treatments and have no other option than enucleation and/or EBR, to preserve functional vision and to limit general and ocular toxicity.

Primary objectives

A. To reduce the incidence of retinal toxicity in IVitC treatment while retaining similar efficacy of tumor control, in vitreous relapse.

B. To reduce further relapse by IAC with melphalan+topotecan compared to IAC with melphalan only in patients not having received prior IAC and presenting retinal / diffuse subretinal relapse.

The primary outcome, on which the sample size calculation is based, is the rate of retinal toxicity following IVitC treatment with melphalan as compared to topotecan. Currently a retinal toxicity rate of 40% is reported with melphalan. Topotecan is reportedly less toxic and the investigators expect a retinal toxicity of 10% or less. To have 90% power of detecting a reduction of 30% in retinal toxicity at the 5% level of significance, 43 patients are required in each arm. Allowing for a 5% drop out rate per year for 3 years, the investigators estimate that 50 patients are required in each of arm of this study. Concerning the second primary objective the investigators postulate that the eye salvage rate can be increased by adding topotecan to melphalan from overall 67% to 84% at 2 years. A randomized 2:1 (arm with association Topotecan-Melphalan and arm with Melphalan only, respectively) non comparative phase II will be performed. In the Topotecan and Melphalan arm, 67% (p0) or less of eye salvage rate is considered as ineffective, 84% (p1) as active. 64 patients will be included in the Topotecan and Melphalan arm, with a type one error of 7% and a type two error of 5%.

ELIGIBILITY:
Inclusion Criteria:

1. Eye with recurrent Rb clinically defined as one or the combination of the following:

   * vitreous recurrence only
   * retinal / diffuse subretinal relapse only not amenable to focal treatment such as thermotherapy, cryotherapy or plaque
   * combined vitreous and retinal/diffuse subretinal relapse
2. Minimally required interval between study entry and time of the last treatment: 2 months (with a monthly follow-up), except for small retinal / subretinal tumors treated focally, not related to the current relapse
3. Photographic documentation of fundus at study entry
4. Registration into the study and start of treatment must occur no later than 14 days after diagnosis of recurrence
5. Mandatory ultrasound biomicroscopy (UBM) at 35 or 50 MHz in case of opaque media or insufficient pupillary dilatation for evaluation of the posterior chamber / pars plana
6. Age ≥3 months and < 11 years (10.99)
7. Weight ≥5 kg (in case of IAC eligibility or sequential IVitC/IAC eligibility)
8. Possibility of follow-up until at least 2 years after end of current relapse treatment
9. Written informed consent by parents or legal representative before enrolment

Exclusion Criteria:

1. Relapse with any uveal involvement and/or anterior chamber involvement
2. Indication for another treatment option according to investigator's judgement
3. Clinical/MRI signs of extraocular disease, including metastatic disease
4. Inadequate organ function (in case of IAC or sequential IVitC / IAC eligibility):

   * absolute neutrophils count <0.5 G/l
   * thrombocytes count <100 G/l
   * creatinine above normal value for age
   * ALAT more than 2x above upper normal limit
   * bilirubin above upper normal limit
5. Other (simultaneous) malignancies
6. Contraindication or known hypersensitivity to study drugs
7. Severe concomitant diseases (e.g. immune deficiency syndrome)
8. Current or recent (within 30 days prior to date of written informed consent) treatment with another investigational drug or participation in another interventional clinical trial

Ages: 3 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Rate of retinal toxicity of intravitreous administration of melphalan versus topotecan assessed by CTCAE v5.0 | at 1 month after treatment completion
  parameters: salt and pepper retinopathy, choroidopathy, number of injections until toxicity
Relapse rate after IAC by melphalan only and IAC by melphalan + topotecan | at 2 years of follow-up
  parameter: eye retention rate

SECONDARY OUTCOMES:
Efficacy of intravitreous topotecan compared to intravitreous melphalan (number of injections to tumor clearance in vitreous) | at 3 or 6 months after last intravitreous injection
  Parameter: number of injections to tumor clearance in vitreous
Ocular survival (eye salvage rate) | at 2 years since study entry
  parameters: enucleation and EBR
Number of participants with ocular (non retinal) and systemic toxicity assessed by CTCAE v5.0 | Weekly (IVitC) or monthly (IAC) during treatment, at end of treatment (1 month after last injection), at 6, 12 and 24 months, yearly until 60 months
  parameter: number of participants
Quality of vision assessed by visual acuity | at 5 years of age
  parameters: Logmar values
Incidence of early (within 1 month), intermediate (2-12 months) and late (> 12 months) ocular and systemic general adverse events during regular ophthalmological and clinical examinationassessed by CTCAE v5.0 | Weekly (IVitC) or monthly (IAC) during treatment, at end of treatment (1 month after last injection), at 6, 12 and 24 months, yearly until 60 months
  parameter: incidence
Quantification of the cumulative radiation exposure during the IAC procedures by routinely used devices (sub-study limited to Lausanne) by B three thermoluminescent dosimeters | at 1 month after the last IAC
  parameter: B three thermoluminescent dosimeters
Incidence of the occurrence of secondary malignancies and/or metastases and long term sequelae | during a follow-up of at least 10 years
  parameter: incidence

CONTACTS AND LOCATIONS:
Overall Officials: Maja Beck Popovic, Prof, Study Director — University of Lausanne Hospitals
Locations (1):
- CHUV Lausanne University Hospital, Lausanne, Switzerland